CLINICAL TRIAL: NCT02829281
Title: Intra-articular Botulinum Toxin Type A Versus Corticosteroids: a Clinical Trial in Osteoarthritis of Knees
Brief Title: Intra-articular Botox Type A Versus Corticosteroids in Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Jamille Godoy Mendes, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP UNIFESP - 319915
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; Intra-articular injection; Botulinum Toxin Type A; Corticosteroid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Botulinum Toxins, Type A; triamcinolone hexacetonide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Botulinum toxin group (Experimental): Patients will receive a intervention with joint injection of 100 units of botulinum toxin
  Interventions: Drug: Botulinum Toxin Type A
- Corticosteroid group (Active Comparator): Patients will receive a intervention with joint injection of 40mg of triamcinolone hexacetonide (corticosteroid)
  Interventions: Drug: Triamcinolone hexacetonide
- Saline Group (Placebo Comparator): Patients will receive a joint injection of 2ml of normal saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Joint injection of Botulinum Toxin Type A
  Arms: Botulinum toxin group
Drug: Triamcinolone hexacetonide — Joint injection of triamcinolone hexacetonide
  Arms: Corticosteroid group
Drug: Saline — Joint injection of Saline
  Arms: Saline Group

SUMMARY:
Introduction: Osteoarthritis of the knee is a very common disease. However there are few treatment options for these patients. Botulinum toxin type A is an option for chronic pain. If the investigators prove effectiveness of its use for intra-articular analgesia, Botulinum toxin type A can be useful for treat these patients.

Objective: Compare the effectiveness of the use of intra-articular corticosteroid versus Botulinum toxin type A in the treatment of patients with knee osteoarthritis.

Methods: A prospective controlled randomized double blind studied with three groups (n = 35 each group) of patients with symptomatic osteoarthritis of the knees receive intra-articular medication in a single moment will be undertaken. The three groups will be: Botulinum toxin type A Group: patients who receive 100 units of botulinum toxin; hexacetonide of triamcinolone Group: patients who receive 40mg of triamcinolone hexacetonide, and saline group: patients who receive 2ml of normal saline. Patients will be assessed by evaluators " blind " in 4 times during 12 weeks of follow-up with clinical assessment instruments (pain, quality of life questionnaire as short form 36 questionnaire) , functional ( WOMAC questionnaire) , and ultrasound (quantitative and semi quantitative measure of synovial hypertrophy and semi quantitative Power Doppler ) .The following statistical tests will be used : Student's t test, Mann - Whitney , chi- square test and ANOVA for repeated measures . Will be considered as statistical significance the difference of 5 %.

ELIGIBILITY:
Inclusion Criteria:

* age above 50 years
* diagnose of knee osteoarthritis using clinics and radiographic criteria
* pain for more than 6 months
* analogic visual scale among 4 to 8
* patients who agree to sign informed consent

Exclusion Criteria:

* secondary osteoarthritis
* skin lesion
* use of intraarticular corticosteroid in the last 3 months
* use of oral corticosteroid in the last 30 days
* Kellgren Lawrence I or IV
* inflammatory arthritis
* neuromuscular disease
* use of aminoglycoside antibiotics
* metalic prosthesis in knee
* peripheric neuropathy
* serious cardiovascular or pulmonary disease
* serious disorder of coagulation
* pregnancy or breastfeeding
* infections
* use of wheelchair

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes on Pain | Baseline, after 4, 8 and 12 weeks
  Evaluated using the visual analogue scale

SECONDARY OUTCOMES:
Changes on Ultrasound parameters | Baseline, after 4, 8 and 12 weeks
  quantitative and semi quantitative measure of synovial hypertrophy and semi quantitative Power Doppler
Changes on quality of life | Baseline, after 4, 8 and 12 weeks
  Evaluated using the Short form 36 questionnaire
Changes on function | Baseline, after 4, 8 and 12 weeks
  Evaluated using the WOMAC questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil